CLINICAL TRIAL: NCT04734665
Title: A Single-arm Phase II Study of Niraparib and Bevacizumab Maintenance Therapy in Platinum-sensitive Recurrent Ovarian Cancer Patients Previously Treated With a PARP Inhibitor
Brief Title: Niraparib and Bevacizumab Maintenance Therapy in Platinum-sensitive Recurrent Ovarian Cancer Patients Previously Treated With a PARP Inhibitor
Acronym: NIRVANA-R
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-0076
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Platinum-sensitive Recurrent Ovarian Cancer Patients Previously Treated With a PARP Inhibitor
Keywords: ovarian cancer, Platinum-sensitive, PARP inhibitor
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): Platinum-sensitive recurrent ovarian cancer patients previously treated with a PARP inhibitor, Non-mucinous
  Interventions: Drug: Niraparib-Bevacizumab

INTERVENTIONS:
Drug: Niraparib-Bevacizumab — Niraparib 200mg or 300mg (once daily[QD]) Bevacizumab 15mg/kg every 3 weeks (Q3W)
  *The recommended starting dosage of niraparib is 200mg QD. For patients who weigh ≥77 kg and have baseline platelet count ≥150,000/μL, the recommended starting dosage is 300 mg QD.

SUMMARY:
This study is phase II, open label, clinical trial to determine the efficacy of Niraparib re-treatment with Bevacizumab of assessment progression-free survival(6 months PFS rate) with platinum-sensitive recurrent ovarian cancer patients previously treated with a PARP inhibitor.

DETAILED DESCRIPTION:
This is a Phase II, open-label, non-randomized, multi-center study assessing the efficacy and safety of Niraparib re-treatment with Bevacizumab of assessment progression-free survival(6 months PFS rate) with platinum-sensitive recurrent ovarian cancer patients previously treated with a PARP inhibitor The study will assess the effectiveness of progression-free survival(6 months PFS rate) as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. The subject will be treated to until disease progression as below:

* Niraparib 200mg or 300mg (once daily[QD])*
* Bevacizumab 15mg/kg every 3 weeks (Q3W)

  * The recommended starting dosage of niraparib is 200mg QD. For patients who weigh ≥77 kg and have baseline platelet count ≥150,000/μL, the recommended starting dosage is 300 mg QD.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has histologically confirmed diagnosis of high-grade predominantly serous, endometrioid, carcinosarcoma, mixed mullerian with high-grade serous component, clear cell, or low-grade serous OC, primary peritoneal cancer, or fallopian tube cancer will be enrolled in this study (only up to 4 patients with clear cell carcinoma will be included and mucinous carcinoma will not be included).
2. Participant has received at least 2 previous courses of platinum-containing therapy, and has disease that was considered platinum sensitive following the penultimate (next to last) platinum course (more than 12 months' period between penultimate platinum regimen and progression of disease) Note: The last platinum regimen does not necessarily have to immediately follow the next to last (penultimate) platinum regimen. For example, if a patient received a non-platinum regimen between the penultimate platinum regimen and last platinum regimen, they could be eligible, so long as they meet all entry criteria.
3. Participant has responded to last the platinum regimen (complete or partial response), remains in response and is enrolled on study within 8 weeks of completion of the last platinum regimen
4. Participant had prior treatment with PARP inhibitor
5. Participant is able to provide a newly obtained core or excisional biopsy of a tumor lesion for prospective testing of BRCA 1/2 and PD-L1 status prior to enrollment
6. Female participants who are at least 20 years of age on the day of signing informed consent with
7. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, as assessed within 10 days prior to enrollment.

   Female participants:
8. A female participant is eligible to participate if she is not pregnant (see Appendix 2), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 2 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 2 during the treatment period and for at least 120 days following the last dose of niraparib and at least 210 days following the last dose of chemotherapy or bevacizumab.

   Informed Consent
9. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial. The participant may also provide consent for future biomedical research; however, the participant may participate in the main study without participating in future biomedical research.
10. Participant has adequate organ function as defined in the following contents; all screening laboratory tests should be performed within 10 days prior to the start of study treatment.

    * Absolute neutrophil count (ANC) ≥1500/µL
    * Platelets ≥100 000/µL
    * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La
    * Creatinine OR Measured or calculated creatinine clearance(GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
    * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
    * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
    * International normalized ratio (INR) OR prothrombin time (PT), Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

1. Participant has mucinous, germ cell, or borderline tumor of the ovary.
2. Participant has a history of non-infectious pneumonitis that required treatment with steroids or currently has pneumonitis
3. Participant either has myelodysplastic syndrome (MDS)/ acute myeloid leukemia (AML) or has features suggestive of MDS/AML.
4. Participant has a known additional malignancy that is progressing or has required active treatment within the past 2 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ, endometrial carinoma) that have undergone potentially curative therapy are not excluded.

   Note: Participants with synchronous primary endometrial cancer or a past history of primary endometrial cancer that met the following conditions are not excluded: Stage not greater than IA: no more than superficial myometrial invasion.
5. Drainage of ascites during last 2 cycles of last chemotherapy.
6. Palliative radiotherapy within 1 week encompassing >20% of the bone marrow.
7. Persistent > grade 2 toxicity from prior cancer therapy.
8. Symptomatic uncontrolled brain or leptomeningeal metastases. A scan to confirm the absence of brain metastases is not required. Patients with spinal cord compression may be considered if they have received definitive treatment for this and evidence of clinically stable disease for 28 days.
9. Known hypersensitivity to the components of niraparib.
10. Major surgery within 3 weeks of starting the study or patient has not recovered from any effects of any major surgery.
11. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
12. History or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study treatment, or is not in the best interest of the patient to participate.
13. Immunocompromised patients.
14. Patients with known active hepatic disease (i.e. , Hepatitis B or C).

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 44 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(6 months PFS rate) | 6 months
  To determine the clinical effectiveness of the study treatment assessed using progression free survival(6months) according to RECIST v1.1 criteria (Investigator determined)

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 1year
Time to tumour progression (TTP) | Up to 1year
Time to first subsequent treatment(or death) | The date of first documented first subsequent treatment or date of death, assessed up to 36months
Time to second subsequent treatment | The date of first documented second subsequent treatment assessed up to 36months
progression-free survival | Up to 1year

CONTACTS AND LOCATIONS:
Overall Officials: Jung Yun Lee, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
(Describe the IPD sharing plan, including what IPD are to be shared with other researchers.)

REFERENCES:
- [Derived] Park J, Lim MC, Lee JK, Jeong DH, Kim SI, Choi MC, Kim BG, Lee JY. A single-arm, phase II study of niraparib and bevacizumab maintenance therapy in platinum-sensitive, recurrent ovarian cancer patients previously treated with a PARP inhibitor: Korean Gynecologic Oncology Group (KGOG 3056)/NIRVANA-R trial. J Gynecol Oncol. 2022 Mar;33(2):e12. doi: 10.3802/jgo.2022.33.e12. Epub 2021 Dec 6. PMID 34910393